CLINICAL TRIAL: NCT04897932
Title: An Evaluation of the Usability and Efficacy of a Prototype Handheld Urinal for Adults Who Suffer From Nocturia, Urge, Frequency, and/or Functional Incontinence
Brief Title: Evaluation Trial of Handheld Urinal for Adult Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Binding Sciences Limited (Industry)
Collaborators: Buckinghamshire Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSL BHT IRAS 291714
Record Dates: First submitted 2021-04-16; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adult nocturia (Active Comparator): Use of device over 28 days
  Interventions: Device: RS - WP06
- Adult urge urinary incontinence (Active Comparator): Use of device over 28 days
  Interventions: Device: RS - WP06
- Adult frequency urinary incontinence (Active Comparator): Use of device over 28 days
  Interventions: Device: RS - WP06
- Adult functional incontinence (Active Comparator): Use of device over 28 days
  Interventions: Device: RS - WP06

INTERVENTIONS:
Device: RS - WP06 — Ad hoc use of handheld urinal

SUMMARY:
Usability and efficacy evaluation of a prototype handheld urinal for adult use

DETAILED DESCRIPTION:
28 day usability and efficacy evaluation by 154 adults in domestic settings who suffer one or more of nocturia, urge, frequency or functional incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Suffers from nocturia urge, frequency, or funnctional incontinence

Exclusion Criteria:

* Suffers only from stress UI

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-30 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in fluid intake | 28 days
  Quantitative analysis of levels of daily fluid intake i) when using the device and ii) not using the device.
Change in incidence of falls associated with urinary toileting | 28 days (3 months reported number of falls based on participant's recollection of incidence during that period)
  Quantitative analysis of the number of falls incurred going to and from toilet while using the device over the 28 day study period compared to the number of falls recalled by participants going to and from the toilet during the 3 months prior to the study when not using the device.
  Tool: user diary and questionairre
Change in level of user independence | 28 days
  Quantitative assessment of number of carer interventions required to assist users with urinary toileting when using and not using the device.
  Tool: user diary and questionairre
Levels of user confidence | 28 days
  Qualitative self-assessments, on a three-point scale of "Not at all confident", "Reasonably confident" and "Very confident", by users of their confidence in their ability to manage urinary incontinence when using the device in a range of different orientations.
  Tool: questionairre
Convenience in use | 28 days
  Qualitative self-assessment by users of the convenience in use of the device relative to other continence aids used on a three-point scale: "More convenient", "Neither more nor less convenient", and "Less convenient".
  Tool: questionairre

CONTACTS AND LOCATIONS:
Overall Officials: Piers Clifford, MD, Principal Investigator — Buckinghamshire Healthcare NHS Trust
Locations (1):
- Binding Sciences Limited, Cropredy, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No